CLINICAL TRIAL: NCT03800485
Title: Effects of Inspiratory Muscle Training on Lung Function, Inspiratory Muscle Strength and Trunk Balance in Patients With Stroke in Subacute Phase.
Brief Title: Inspiratory Muscle Training in Patients With Stroke in Subacute Phase.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Virgen de la Arrixaca (Other)
Collaborators: Universidad Católica San Antonio de Murcia (Other); Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, Alicia Tovar Alcaraz, Physical therapist, Hospital Universitario Virgen de la Arrixaca
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-10-4-HCUVA
Record Dates: First submitted 2018-12-17; First posted 2019-01-11 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Stroke Rehabilitation
Keywords: stroke; respiratory muscles; lung; stroke rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: There are two groups, the intervention group and the placebo group.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study is blinded so neither the patient, neither the psysical therapist nor the investigator knows in which group the patient is
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMT-GE (Experimental): the participants will perform a training protocol of the inspiratory muscles during 8 weeks with a load that will increase from the 15% of the maximal inspiratory preassure until the 60% of the maximal inspiratory preassure.
  Interventions: Device: IMT
- IMT-GP (Placebo Comparator): The participants will perform a training protocol of the inspiratory muscles during 8 weeks with a load that will be the 10% of the maximal inspiratory preassure during all the 8 weeks
  Interventions: Device: IMT

INTERVENTIONS:
Device: IMT — A training protocol of the inspiratory muscles that goes from the 15% of the maximal inspiratory muscle preassure until the 60% of the maximal inspiratory muscle preassure during 8 weeks

SUMMARY:
Assess the effect of inspiratory muscle training on lung function, muscle strength and trunk balance in survivors of stroke in the subacute phase of the disease

DETAILED DESCRIPTION:
Assess the effect of inspiratory muscle training on lung function, muscle strength and trunk balance in survivors of stroke in the subacute phase of the disease. The intervention will be done in a group of patients who will be treated in the rehabilitation service at the Virgen de la Arrixaca Hospital. They will train using a threshold IMT device or a Powerbreathe device, to increase their inspiratory muscle strength in addition to a physical therapy treatment. The intervention will last eigtht weeks and the patients will be evaluated at the beginning and at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Sroke 6 months before of the beginning of the study
* Be able to understand simple commands
* Hemiparesis or hemiplegia
* Not have serious cardiopulmonary diseases(COPD,asthma,bronchiectasis)

Exclusion Criteria:

* Associated neurological pathology leading to muscle weakness
* Severe respiratory pathology, pulmonary embolism, presence of tracheostomy cannula,
* intracranial hypertension
* Acute retinal datachment, recent eye surgery
* Impossibility of labial occlusion
* Unstable heart disease, unstable angina, aortic aneurysm
* Recent thoracic or abdominal surgery(6 months)
* Uncontrolled arterial hypertension

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-01-20 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Maximum inspiratory pressure | From the first day of evaluation and at eight weeks of the beginning of the intervention
  The change of the maximum inspiratory pressure from the beginning, at 4 weeks and At 8 weeks
Forzed vital capacity | From the first day of evaluation and at eight weeks of the beginning of the intervention
  The change of the forzed vital capacity from the beginning and at the end of the intervention
Forzed espiratory volume in the first second | From the first day of evaluation and at eight weeks of the beginning of the intervention
  The change of the forzed espiratory volumen in the first second beginning and in the end of the intervention using a spirometer
Voluntary maximum ventilation | From the first day of evaluation and at eight weeks of the beginning of the intervention
  The change of the voluntary maximum ventilation from the beginning and at the end of the intervention using a spirometer
The "Berg balance scale" Test | From the first day of evaluation and at Eight weeks of the beginning of the intervention
  The change of the balance at the beginning and in the end of the intervention using the berg balance scale tool. The máximum value of this scale is 56 points, and the mínimum is 0 points. A higher value represents a better outcome.
The postural assessment scale for stroke patients (PASS )test | From the first day of evaluation and at Eight weeks of the beginning of the intervention
  The change of the balance of the trunk at the beginning and in the end of the intervention using the postural assessment scale for stroke patinents tool. The maximum value of tris scale is 36 points. The minimum is 0 points.Higher values represents a better outcome.
Trunk control test (TCT) | From the first day of evaluation and at Eight weeks of the beginning of the intervention
  The change of the trunk control at the beginning and in the end of the intervention. The maximum value is 100 points, and the minimum 0 points. Higher values represents a better outcome

SECONDARY OUTCOMES:
Quadriceps dynamometry | From the first day of evaluation and at eight weeks of the beginning of the intervention
  The change of the quadriceps´s strength with a hand held dynamometer at the beginning and in the end of the intervention. Higher values represents a better outcome
"Functional ambulatory classificator" Test | From the first day of evaluation and at Eight weeks of the beginning of the intervention
  The change of the walking capacity using the functional ambulatory classificator tool at the beginning and in the end of the intervention. The máximum value is 5 and the mínimum 0. Higher values represents a better outcome
"Functional ambulatory classificator Hospital de Sagunto" Test | From the first day of evaluation and at Eight weeks of the beginning of the intervention
  The change of the walking capacity using the functional ambulatory classificator hospital de sagunto tool at the beginning and ni the end. The máximum value is 5 and the mínimum 0. Higher valúes represents better outcome
SF-36 health survey | From the first day of evaluation and at eight weeks of the beginning of the intervention
  The change of the quality of life related to health with the SF-36 health survey at the beginning and in the end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: MARTHA C LEON GARZON, PhD, Study Director — UNIVERSIDAD SAN ANTONIO DE MURCIA; SILVANA L DE OLIVEIRA SOUSA, PhD, Study Director — Universidad Miguel Hernandez, Elche; ALICIA TOVAR ALCARAZ, Pt, Principal Investigator — Hospital Universitario Virgen de la Arrixaca
Locations (1):
- Alicia Tovar Alcaraz, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data includes the spirometry data

REFERENCES:
- [Result] Messaggi-Sartor M, Guillen-Sola A, Depolo M, Duarte E, Rodriguez DA, Barrera MC, Barreiro E, Escalada F, Orozco-Levi M, Marco E. Inspiratory and expiratory muscle training in subacute stroke: A randomized clinical trial. Neurology. 2015 Aug 18;85(7):564-72. doi: 10.1212/WNL.0000000000001827. Epub 2015 Jul 15. PMID 26180145
- [Result] Sutbeyaz ST, Koseoglu F, Inan L, Coskun O. Respiratory muscle training improves cardiopulmonary function and exercise tolerance in subjects with subacute stroke: a randomized controlled trial. Clin Rehabil. 2010 Mar;24(3):240-50. doi: 10.1177/0269215509358932. Epub 2010 Feb 15. PMID 20156979
- [Result] Kulnik ST, Birring SS, Moxham J, Rafferty GF, Kalra L. Does respiratory muscle training improve cough flow in acute stroke? Pilot randomized controlled trial. Stroke. 2015 Feb;46(2):447-53. doi: 10.1161/STROKEAHA.114.007110. Epub 2014 Dec 11. PMID 25503549
- [Result] Kim CY, Lee JS, Kim HD, Kim IS. Effects of the combination of respiratory muscle training and abdominal drawing-in maneuver on respiratory muscle activity in patients with post-stroke hemiplegia: a pilot randomized controlled trial. Top Stroke Rehabil. 2015 Aug;22(4):262-70. doi: 10.1179/1074935714Z.0000000020. Epub 2015 Feb 18. PMID 26258451
- [Result] Jung KM, Bang DH. Effect of inspiratory muscle training on respiratory capacity and walking ability with subacute stroke patients: a randomized controlled pilot trial. J Phys Ther Sci. 2017 Feb;29(2):336-339. doi: 10.1589/jpts.29.336. Epub 2017 Feb 24. PMID 28265169